CLINICAL TRIAL: NCT02200978
Title: A Multicenter and Randomized Prospective Study for Improving the Outcome of Childhood Acute Promyeloid Leukemia
Brief Title: A Study for Improving the Outcome of Childhood Acute Promyeloid Leukemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: South China Children's Leukemia Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010001
Record Dates: First submitted 2014-02-08; First posted 2014-07-25 (Estimated); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Childhood Acute Promyelocytic Leukemia
MeSH Terms: interventions — Arsenic Trioxide; Tretinoin; Mitoxantrone; Cytarabine; Methotrexate; Mercaptopurine; Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATO and chemotherapy (Active Comparator): Induction:
  ATRA 25mg/m2 d1-CR ≯42 days; ATO 0.16mg/kg d5-CR ≯42 days; mitoxantrone (MA) 10mg/m2 d3, or 7mg/m2 d2-4 (high risk).
  Consolidation 1:
  ATRA 25mg/m2 d1-15; MA 10mg/m2 d1-2; Intrathecal injection (IT)：Ara-C 15mg (age < 1 year), or 20 mg (1-3 years), or 30 mg ( > 3 years), dexamethasone 2mg.
  Consolidation 2:
  ATRA 25mg/m2 d1-15; ATO 0.16mg/kg d1-15; Ara-C 1g/m2 q12h d1-2 (high risk); IT.
  Consolidation 3:
  ATRA 25mg/m2 d1-15; ATO 0.16mg/kg d1-15; MA 10mg/m2 d1; Ara-C 1g/m2 q12h d1-2 (high risk); IT.
  Maintenance:
  ① ATO 0.16mg/kg.d w1-2; ATRA 25mg/m2.d w1-2; MTX 20mg/m2 qw w3-12; 6MP 50mg/m2 qn w3-12. ② ATRA 25mg/m2.d w1-2; MTX 20mg/m2 qw w3-12; 6MP 50mg/m2 qn w3-12. Rotation between ① and ② until the end of maintenance.
  Interventions: Drug: ATO; Drug: ATRA; Drug: mitoxantrone; Drug: Ara-C; Drug: MTX; Drug: 6MP; Other: intrathecal injection
- RIF and chemotherapy (Experimental): Induction:
  ATRA 25mg/m2 d1-CR ≯42 days; RIF 0.135/kg d5-CR ≯42 days; mitoxantrone (MA) 10mg/m2 d3, or 7mg/m2 d2-4 (high risk).
  Consolidation 1:
  ATRA 25mg/m2 d1-15; MA 10mg/m2 d1-2; Intrathecal injection (IT)：Ara-C 15mg (age < 1 year), or 20mg (age 1-3 years), or 30mg (age > 3 years), dexamethasone 2mg.
  Consolidation 2:
  ATRA 25mg/m2 d1-15; RIF 0.135/kg d1-15; Ara-C 1g/m2 q12h d1-2 (high risk); IT.
  Consolidation 3:
  ATRA 25mg/m2 d1-15; RIF 0.135/kg d1-15; MA 10mg/m2 d1; Ara-C 1g/m2 q12h d1-2 (high risk); IT.
  Maintenance:
  ① RIF 0.135/kg.d w1-2; ATRA 25mg/m2.d w1-2; MTX 20mg/m2 qw w3-12; 6MP 50mg/m2 qn w3-12. ② ATRA 25mg/m2.d w1-2; MTX 20mg/m2 qw w3-12; 6MP 50mg/m2 qn w3-12. Rotation between ① and ② until the end of maintenance treatment.
  Interventions: Drug: RIF; Drug: ATRA; Drug: mitoxantrone; Drug: Ara-C; Drug: MTX; Drug: 6MP; Other: intrathecal injection

INTERVENTIONS:
Drug: ATO — Given IV
  Other Names: As2O3; arsenic trioxide
  Arms: ATO and chemotherapy
Drug: RIF — Given orally
  Other Names: Realgar-Indigo naturalis formula
  Arms: RIF and chemotherapy
Drug: ATRA — Given orally
  Other Names: all-trans retinoic acid
Drug: mitoxantrone — Given IV
  Other Names: novantrone
Drug: Ara-C — Given IV
  Other Names: cytarabine; cytosine arabinoside
Drug: MTX — Given orally
  Other Names: methotrexate
Drug: 6MP — Given orally
  Other Names: mercaptopurine
Other: intrathecal injection — Ara-C and dexamethasone
  Other Names: IT

SUMMARY:
Outcome of acute promyelocytic leukemia (APL) has greatly improved since the introduction of all-trans-retinoic acid (ATRA). Treatment with ATRA and anthracycline-based chemotherapy (ATRA + chemotherapy) decreases relapses of the disease as well as early hemorrhagic deaths. Nowadays patients with APL have an event-free survival (EFS) of up to 80%. However, there remains a subset of the patients in whom the disease relapses. Recently, a randomized prospective study showed that the addition of ATO to "ATRA + chemotherapy" treatment protocol had a significantly higher EFS in patients with APL than those treated with "ATRA + chemotherapy" protocol. The patients treated with "ATO + ATRA + chemotherapy" had a five years EFS of 89.2%. Moreover, a recent study showed that Indigo naturalis formula (RIF), a traditional Chinese medicine with tetraarsenic tetrasulfide (As4S4), indirubin, and tanshinone IIA as major active ingredients, yielded synergy in the treatment of a murine APL model in vivo and in the induction of APL cell differentiation in vitro . It is about 20 years since RIF was used to treat ALP in China. Clinical studies showed that this agent was effective against APL. Compared to ATO, RIF is relatively inexpensive and can be taken orally, resulting in reducing the number of hospital days and the treatment cost. However, there is no report comparing treatment outcomes of "ATO + ATRA + chemotherapy" and "RIF + ATRA + chemotherapy" protocols in children with APL so far. For this purpose, therefore, investigators are going to conduct a multicenter and randomized prospective study in children with APL.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and efficacy of "ATO/RIF + ATRA + less intensive chemotherapy" protocol in children with acute promyelocytic leukemia (APL).
* Compare the safety，efficacy and treatment cost of "RIF + ATRA + less intensive chemotherapy" with "ATO + ATRA + less intensive chemotherapy" protocol in children with APL. Determine if ATO can be substituted by RIF.

OUTLINE: This is a multicenter and randomized prospective study.

PROJECTED ACCRUAL: A total of 162 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 16 years old with newly diagnosed PML-RARa positive acute promyelocytic leukemia.

Exclusion Criteria:

* Patients who have coma, convulsion or paralysis due to intracranial hemorrhage or central nervous system leukemia at diagnosis.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2011-09; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
event-free survival | 5 years

SECONDARY OUTCOMES:
hospitalization cost | 2 years
  The cost mainly includes the fees of hospital bed, drugs, therapies and blood products. Time frame: from the beginning of induction therapy to the end of maintenance treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Qun Luo, professor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shen ZX, Shi ZZ, Fang J, Gu BW, Li JM, Zhu YM, Shi JY, Zheng PZ, Yan H, Liu YF, Chen Y, Shen Y, Wu W, Tang W, Waxman S, De The H, Wang ZY, Chen SJ, Chen Z. All-trans retinoic acid/As2O3 combination yields a high quality remission and survival in newly diagnosed acute promyelocytic leukemia. Proc Natl Acad Sci U S A. 2004 Apr 13;101(15):5328-35. doi: 10.1073/pnas.0400053101. Epub 2004 Mar 24. PMID 15044693
- [Background] Hu J, Liu YF, Wu CF, Xu F, Shen ZX, Zhu YM, Li JM, Tang W, Zhao WL, Wu W, Sun HP, Chen QS, Chen B, Zhou GB, Zelent A, Waxman S, Wang ZY, Chen SJ, Chen Z. Long-term efficacy and safety of all-trans retinoic acid/arsenic trioxide-based therapy in newly diagnosed acute promyelocytic leukemia. Proc Natl Acad Sci U S A. 2009 Mar 3;106(9):3342-7. doi: 10.1073/pnas.0813280106. Epub 2009 Feb 18. PMID 19225113
- [Background] Wang L, Zhou GB, Liu P, Song JH, Liang Y, Yan XJ, Xu F, Wang BS, Mao JH, Shen ZX, Chen SJ, Chen Z. Dissection of mechanisms of Chinese medicinal formula Realgar-Indigo naturalis as an effective treatment for promyelocytic leukemia. Proc Natl Acad Sci U S A. 2008 Mar 25;105(12):4826-31. doi: 10.1073/pnas.0712365105. Epub 2008 Mar 14. PMID 18344322
- [Background] Xiang Y, Wang XB, Sun SJ, Guo AX, Wei AH, Cheng YB, Huang SL. [Compound huangdai tablet as induction therapy for 193 patients with acute promyelocytic leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2009 Jul;30(7):440-2. Chinese. PMID 19954593
- [Background] Luo XQ, Ke ZY, Huang LB, Guan XQ, Zhang YC, Zhang XL. Improved outcome for Chinese children with acute promyelocytic leukemia: a comparison of two protocols. Pediatr Blood Cancer. 2009 Sep;53(3):325-8. doi: 10.1002/pbc.22042. PMID 19422024
- [Derived] Fan Z, Yang LC, Chen YQ, Wan WQ, Zhou DH, Mai HR, Li WL, Yang LH, Lan HK, Chen HQ, Guo BY, Zhen ZJ, Liu RY, Chen GH, Feng XQ, Liang C, Wang LN, Yu-Li, Luo JS, Huang DP, Luo XQ, Li B, Huang LB, Zhang XL, Tang YL. Prognostic significance of MRD and its correlation with arsenic concentration in pediatric acute promyelocytic leukemia: a retrospective study by SCCLG-APL group. Ther Adv Hematol. 2025 Jan 7;16:20406207241311774. doi: 10.1177/20406207241311774. eCollection 2025. PMID 39781038
- [Derived] Liao LH, Chen YQ, Huang DP, Wang LN, Ye ZL, Yang LH, Mai HR, Li Y, Liang C, Luo JS, Wang LN, Luo XQ, Tang YL, Zhang XL, Huang LB. The comparison of plasma arsenic concentration and urinary arsenic excretion during treatment with Realgar-Indigo naturalis formula and arsenic trioxide in children with acute promyelocytic leukemia. Cancer Chemother Pharmacol. 2022 Jul;90(1):45-52. doi: 10.1007/s00280-022-04449-9. Epub 2022 Jun 27. PMID 35760920